CLINICAL TRIAL: NCT05212454
Title: Efficacy and Safety of Supplement Adjuvant Capecitabine in Postoperative Hormone Receptor (HR)-Positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative High-risk Breast Cancer Patients: a Multicenter, Single-arm Clinical Trial
Brief Title: Efficacy of Supplement Adjuvant Capecitabine in HR+/HER2- Breast Cancer Patients With High Risks
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Wei Tian, Vice Director of Department of Breast Surgery and Oncology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1116
Record Dates: First submitted 2022-01-15; First posted 2022-01-28 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Chemotherapy Effect
Keywords: breast cancer; HR positive HER2 negative; high-risk factors; capecitabine; adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capecitabine group (Experimental): All enrolled cases should be given standard chemotherapy, radiotherapy and endocrine therapy according to the Chinese Society of Clinical Oncology (CSCO) guidelines for the treatment of breast cancer, with the specific regimen decided by the doctor according to the condition. After the completion of standard chemotherapy, capecitabine 1250mg/m2 should be given orally twice a day for 2 weeks of the 3-week treatment course, and the total duration of treatment is 8 courses, which can be given simultaneously with radiotherapy and endocrine therapy. Premenopausal patients may use ovarian suppressants as needed.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — capecitabine, 0.5g per pill, given 1250mg/m2 twice a day for 2 weeks of the 3-week treatment course. The total duration of treatment is 8 courses.

SUMMARY:
According to the latest data from the World Health Organization's International Agency for Research on Cancer (IARC) for 2020, breast cancer has been the most prevalent cancer with 2.26 million new cases. Among Chinese breast cancer patients, approximately 60% are hormone receptor (HR) positive, and 80% have early-stage breast cancer. For HR-positive, human epidermal growth factor receptor-2 (HER2) negative breast cancer patients, the first peak of recurrence is about 2-3 years after surgery, especially for patients with high-risk clinical and/or pathological features. Therefore, adjuvant therapy is essential to reduce recurrence during this period.

Capecitabine is an anti-metabolite fluoropyrimidine deoxynucleoside carbamate that can be converted to fluorouracil (5-Fu) in vivo. Studies have shown that patients with HR-positive HER2-negative breast cancer with high-risk factors may benefit from postoperative adjuvant capecitabine therapy as well as patients with triple-negative breast cancer. Therefore, we assumed that additional capecitabine may reduce the reccurence of breast cancer in patients with high-risk factors.

This trial is an open, single-arm clinical trial designed to investigate the effect of additional adjuvant capecitabine therapy on recurrence and survival in HR-positive HER2-negative breast cancer patients with high-risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18-70 years.
* Completed radical breast cancer surgery with confirmed pathology suggested primary invasive breast adenocarcinoma, ER and/or PR positive (defined as positive cells >1%) and HER2 negative (defined as HER2 immunohistochemistry 2+ or less and FISH negative).
* Definition of high-risk factors: 4 or more positive axillary lymph nodes; 1-3 positive axillary lymph nodes with primary tumor ≥ 5 cm or histologic grade 3 or ki67 ≥ 20%; or residual lesions despite neoadjuvant chemotherapy.
* No prior treatment for present breast cancer onset.
* ECOG physical status score 0 to 1
* Hematological examination before treatment should meet: white blood cell count (WBC) ≥ 4.0×10^9/L, neutrophil count (ANC) ≥ 1.5×10^9/L, platelet count (PLT) ≥ 100×10^9/L; hemoglobin (Hb) ≥ 90g/L; AST (sGOT), ALT (sGPT) ≤ 1.5 times the normal value upper limit, creatinine ≤ 1.5 times the upper limit of normal value, total bilirubin ≤ 1.5 times the upper limit of normal value.
* No serious impairment of heart, liver, kidney and other important organ functions.

Exclusion Criteria:

* Unwilling or unable to use an acceptable method of contraception for up to and including 8 weeks after the final dose of the test drug.
* Women during pregnancy and breastfeeding after pregnancy.
* Women with proven distant metastases of breast cancer.
* Patients with proven sensory or motor nerve disease.
* Definite cardiovascular disease, severe co-morbidity or active infection, including known HIV infection.
* Patients who need long-term anticoagulant drugs for cardiovascular or thrombotic diseases.
* History of other tumors.
* Allergic to the study drug or its excipients, etc.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  defined as the time from randomization to recurrence in situ, metastasis, contralateral breast cancer, second primary cancer, and all-cause death.

SECONDARY OUTCOMES:
overall survival | 5 years
  defined as the time from randomizeation to all-cause death
invasive disease free survival | 5 years
  Defined as time from randomization to local or distant recurrence of invasive cancer

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang Univercity School of Medicine, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan L, Strasser-Weippl K, Li JJ, St Louis J, Finkelstein DM, Yu KD, Chen WQ, Shao ZM, Goss PE. Breast cancer in China. Lancet Oncol. 2014 Jun;15(7):e279-89. doi: 10.1016/S1470-2045(13)70567-9. PMID 24872111
- [Background] Yin W, Di G, Zhou L, Lu J, Liu G, Wu J, Shen K, Han Q, Shen Z, Shao Z. Time-varying pattern of recurrence risk for Chinese breast cancer patients. Breast Cancer Res Treat. 2009 Apr;114(3):527-35. doi: 10.1007/s10549-008-0022-5. Epub 2008 Apr 19. PMID 18425576
- [Background] Mamounas EP, Tang G, Paik S, Baehner FL, Liu Q, Jeong JH, Kim SR, Butler SM, Jamshidian F, Cherbavaz DB, Sing AP, Shak S, Julian TB, Lembersky BC, Lawrence Wickerham D, Costantino JP, Wolmark N. 21-Gene Recurrence Score for prognosis and prediction of taxane benefit after adjuvant chemotherapy plus endocrine therapy: results from NSABP B-28/NRG Oncology. Breast Cancer Res Treat. 2018 Feb;168(1):69-77. doi: 10.1007/s10549-017-4550-8. Epub 2017 Nov 11. PMID 29128898
- [Background] Natori A, Ethier JL, Amir E, Cescon DW. Capecitabine in early breast cancer: A meta-analysis of randomised controlled trials. Eur J Cancer. 2017 May;77:40-47. doi: 10.1016/j.ejca.2017.02.024. Epub 2017 Mar 27. PMID 28355581
- [Background] Walko CM, Lindley C. Capecitabine: a review. Clin Ther. 2005 Jan;27(1):23-44. doi: 10.1016/j.clinthera.2005.01.005. PMID 15763604
- [Background] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Background] Joensuu H, Kellokumpu-Lehtinen PL, Huovinen R, Jukkola-Vuorinen A, Tanner M, Kokko R, Ahlgren J, Auvinen P, Paija O, Helle L, Villman K, Nyandoto P, Nilsson G, Pajunen M, Asola R, Poikonen P, Leinonen M, Kataja V, Bono P, Lindman H. Adjuvant capecitabine, docetaxel, cyclophosphamide, and epirubicin for early breast cancer: final analysis of the randomized FinXX trial. J Clin Oncol. 2012 Jan 1;30(1):11-8. doi: 10.1200/JCO.2011.35.4639. Epub 2011 Nov 21. PMID 22105826